CLINICAL TRIAL: NCT02435771
Title: Efficacy Of Ergocalciferol In Adults According To BMI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: failed to meet enrollment goals
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 359128-8
Record Dates: First submitted 2013-05-21; First posted 2015-05-06 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Obesity; Vitamin D Deficiency
MeSH Terms: conditions — Obesity; Vitamin D Deficiency | interventions — Ergocalciferols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BMI <25 (Experimental): Normal BMI
  Interventions: Drug: Ergocalciferols
- BMI 25-35 (Experimental): Overweight and obese by BMI
  Interventions: Drug: Ergocalciferols
- BMI >35 (Experimental): Obese by BMI
  Interventions: Drug: Ergocalciferols

INTERVENTIONS:
Drug: Ergocalciferols — Treatment 1- 400,000 IU
Drug: Ergocalciferols — Treatment 2- 800,000 IU

SUMMARY:
Vitamin D insufficiency is an increasing trend in the United States. According to the NHANES data collection there was a near doubling of patients with vitamin D deficiency in 10 years. Vitamin D deficiency is associated with several adverse outcomes such as increased fractures, certain microbial diseases, cardiovascular diseases, and metabolic dysfunction. The increasing prevalence of vitamin D deficiency has been attributed to the increasing prevalence of obesity. Several studies have shown that obese patients have lower 25-OH vitamin D (25-OHD) levels compared to nonobese patients and obese patients require more vitamin D compared to nonobese patients. The most commonly prescribed medication to replete vitamin D deficiency is oral ergocalciferol. To date, no prospective trials have been published to evaluate a standard protocol in the treatment of vitamin D insufficiency in adults.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects have to be between the ages of 18 to 65 with a serum 25OHD level less than 20 ng/ml.

Exclusion Criteria:

* Participants will be excluded if they have any of the following:

  1. Due to the inaccuracies of BMI in patients with increased muscle mass, in group with a BMI 25-35: men with a waist circumference < 90 cm ; women < 80 cm
  2. Chronic liver disease defined by any clinical or a history of serum AST or ALT > 2 times ULN
  3. Kidney disease defined as a GFR <60 ml/min
  4. Sarcoidosis
  5. Any known malignancy
  6. Known malabsorption disorder to include inflammatory bowel disease, celiac disease, cystic fibrosis, history of gastric bypass
  7. Primary hyperparathyroidism or hypercalcemia,
  8. Patients that are pregnant or considering pregnancy.
  9. Patients taking certain medications such as glucocorticoids, anti-seizure medications such has phenobarbital or phenytoin or patients taking antiviral medications for HIV as these are known to cause vitamin D deficiency
  10. Individuals excluded from having a DXA scan

Study participants will be excluded from having a DXA scan if any of the following:

1. Any amputation of a extremity including toes
2. If they have a pacemaker, automatic defibrillator, coronary stents or metal suture material in the heart
3. If they have artificial joints, pins, plate or any other type of metal objects
4. If they have received contrast material such as barium in the past 7 days
5. If they have had a nuclear medicine study in the past 3 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-07; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
serum 25-hydroxy-vitamin D level | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alicia L Warnock, MD, Principal Investigator — WRNMMC-B; Patrick W Clyde, MD, Study Director — WRNMMC-B; Vinh Mai, MD, Study Chair — WRNMMC-B; Verna Parchment, Study Chair — WRNMMC-B
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States